CLINICAL TRIAL: NCT01099722
Title: Assessment of the Efficacy and Safety of FlutiForm® pMDI 125/5 µg (2 Puffs Bid) Versus Symbicort® Turbohaler® 200/6 µg (2 Puffs Bid) in Adolescent and Adult Subjects With Moderate to Severe Persistent, Reversible Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FLT3507; 2009-017223-25
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: moderate to severe persistent reversible asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaler (Active Comparator)
  Interventions: Drug: Flutiform; Drug: Symbicort Turbohaler
- inhaler (Active Comparator): Symbicort
  Interventions: Drug: Symbicort Turbohaler

INTERVENTIONS:
Drug: Flutiform — inhaler 2 puffs bd daily
Drug: Symbicort Turbohaler — 2 puffs bd daily

SUMMARY:
A comparator study to assess safety and efficacy of Flutiform® compared with symbicort turbohaler in asthma patients with moderate to severe persistent, reversible asthma.

DETAILED DESCRIPTION:
This is a study involving a 2-4 week run-in phase followed by a 12 week double blind treatment phase. During the run-in phase, subjects receive Flixotide®. In the treatment phase subjects will be randomised to one of the two treatment groups and will receive either FlutiForm® and placebo inhaler for symbicort® turbohaler® or symbicort® turbohaler® and placebo inhaler for Flutiform ® . Efficacy will be assessed by lung function tests, asthma symptoms, sleep disturbance due to asthma and rescue medication use. Safety will be assessed by adverse events, lab tests, ECGs and vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 12 years old
2. Female subjects less than 1 year post-menopausal must have a negative urine pregnancy test recorded at the screening visit prior to the first dose of study medication, be non-lactating, & willing to use adequate & highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently & correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner.
3. Known history of moderate to severe persistent, reversible asthma for ≥ 6 months prior to the Screening Visit characterised by:

   Treatment with an inhaled corticosteroid (ICS) at a dose of 250 - 1000 µg fluticasone or equivalent OR Treatment wth ICS at a dose of 200-500 µg fluticasone or equivalent in combination with a Long Acting β2-Agonist (LABA).
4. Demonstrated a FEV1 of ≥ 50% to ≤ 80% for predicted normal values (Quanjer et al., 1993 (adults), & 1995 (adolescents)) during the Screening Period (Visit 1 or Visit 2) following appropriate withholding of asthma medications (if applicable).

   * No β2-agonist use on day of testing
   * No use of inhaled combination asthma therapy on day of testing.
   * Inhaled corticosteroids are allowed on day of testing.
5. Documented reversibility of ≥ 15% in FEV1 at visit 1 or visit 2.
6. Demonstrated satisfactory technique in the use of the study medications i.e. pMDI and Dry Powder Inhaler (DPI) devices.
7. Willing & able to enter information in the electronic diary & attend all study visits.
8. Willing & able to substitute study medication for their pre study prescribed asthma medication for the duration of the study.
9. Written informed consent obtained. Inclusion criteria required following run-in: Subject has used rescue medication for at least 3 days & had at least 1 night with sleep disturbance (i.e., sleep disturbance score of ≥ 1) during the last 7 days of the run in period,OR subject has used rescue medication for at least 3 days & had at least 3 days with asthma symptoms (i.e., a symptom score of ≥ 1) during the last 7 days of the run-in period.

Exclusion criteria:

1. Near fatal or life-threatening (including intubation) asthma within the past year.
2. Hospitalisation or an emergency visit for asthma within the 4 weeks before the Screening Visit.
3. Known history of systemic (injectable or oral) corticosteroid medication use within 1 month of the Screening Visit.
4. Known history of omalizumab use within the past 6 months.
5. Current evidence or known history of any clinically significant disease or abnormality including uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia. 'Clinically significant' is defined as any disease that, in the opinion of the Investigator, would put the subject at risk through study participation, or which would affect the outcome of the study.
6. In the investigator's opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to the Screening Visit.
7. Significant, non-reversible, active pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, tuberculosis).
8. Known Human Immunodeficiency Virus (HIV)-positive status.
9. Subject has a smoking history equivalent to "10 pack years" (i.e., at least 1 pack of 20 cigarettes/day for 10 years or 10 packs/day for 1 year, etc.).
10. Current smoking history within 12 months prior to the Screening Visit.
11. Current evidence or known history of alcohol and/or substance abuse within 12 months prior to the Screening Visit.
12. Subject has taken B-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within the past week.
13. Current use of medications other than those allowed in the protocol that will have an effect on bronchospasm &/or pulmonary function.
14. Current evidence or known history of hypersensitivity or idiosyncratic reaction to test medications or components.
15. Subject has received an investigational drug within 30 days of the Screening Visit (12 weeks if an oral or injectable steroid).
16. Subject is currently participating in a clinical study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2010-04; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
non-inferiority in the efficacy of FlutiForm® | baseline to the end of the 12 week treatment
  To show non-inferiority in the efficacy of FlutiForm® pMDI 125/5 µg (2 puffs bid) vs Symbicort® Turbohaler® 200/6 µg (2 puffs bid), based on the mean change in the pre morning dose value of forced expiratory volume in the first second (FEV1) from baseline (end of run-in period) to the end of the 12 week treatment period.

SECONDARY OUTCOMES:
Additional efficacy and safety assessments
  efficacy assessments include patient centered outcome assessments such as asthma quality of life questionnaire, subject's assessment of study medication, amount of rescue medication use, asthma symptom scores, sleep disturbance due to asthma, discontinuations due to lack of efficacy, compliance with study medication use & asthma exacerbations. Post dose FEV1, peak expiratory flow rates & other lung function parameters.
  Safety assessments include incidence & type of spontaneously reported adverse events, vital signs, laboratory tests and 12-lead ECGs.

CONTACTS AND LOCATIONS:
Locations (5):
- Sofia, Bulgaria
- Csongrád Megyei Önkormányzat Mellkasi Betegségek Szakkórháza Tüdőgondozó Intézet, Szeged, Hungary
- Indore, India
- Krakow, Poland
- Brasov, Romania

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: Results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT3507